CLINICAL TRIAL: NCT03639012
Title: Observational Outcomes in Paediatric Patients Who Receive Preoperative Carbohydrate Loading for Adenoidectomy and Tonsillectomy, a Randomised Control Trial
Brief Title: Outcomes of Carbohydrate Loading Paediatric Patients Preoperatively for Tonsillectomy and Adenoidectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Jessica Gray (Other)
Responsible Party: Sponsor-Investigator, Jessica Gray, Principal Investigator Jessica Gray, IWK Health Centre
Organization: IWK Health Centre (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Paeds ERAS for T&A
Record Dates: First submitted 2018-07-11; First posted 2018-08-20 (Actual); Last update posted 2018-08-21 (Actual); Status verified 2018-08

CONDITIONS: Postoperative Pain; Postoperative Nausea; Satisfaction; Sleep; Postoperative Complications
MeSH Terms: conditions — Pain, Postoperative; Postoperative Nausea and Vomiting; Personal Satisfaction; Postoperative Complications

STUDY DESIGN:
Intervention Model Description: Randomised control trial into 1 of 2 groups
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Carbohydrate loading (Active Comparator): Patients to receive an oral preoperative carbohydrate drink
  Interventions: Dietary Supplement: Carbohydrate drink
- No Carbohydrate loading (No Intervention): Current standard of care

INTERVENTIONS:
Dietary Supplement: Carbohydrate drink — Children randomised to this group will receive a preoperative carbohydrate drink 90-120mins prior to surgery
  Arms: Carbohydrate loading

SUMMARY:
Randomised control trial of 150 paediatric patients aged between 3-8years. One group will receive a preoperative carbohydrate oral drink and the other group will receive current standard care (no drink) prior to undergoing tonsillectomy and/or adenoidectomy.

Outcomes to be reported will be: 1) patient and parent satisfaction; 2) post operative pain score at: recover, 1 hour post op, prior to discharge home and then day 1 postoperatively; 3) PONV rates in recovery, prior to discharge home and again on Day 1 postoperatively; 4) sleep quality night after surgery.

DETAILED DESCRIPTION:
Children undergoing tonsillectomy and/or adenoidectomy will be consented via parents prior to the day of surgery and then randomised to 1 of 2 groups who will either receive the intervention or current standard care. Patients will be recruited from the ENT outpatient clinics in conjunction with the ENT surgeons.

Data collection will be undertaken with the aid of experience research assistants.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing Tonsillectomy and/or adenoidectomy
* consented to undertake preop carbohydrate drink and follow up procedures

Exclusion Criteria:

* Increased risk of aspiration or unable to swallow liquids
* outside age range
* non-consent to undertake treatment or follow up

Ages: 3 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 150 (Estimated)
Dates: Start 2018-09 (Estimated); Primary Completion 2020-02 (Estimated); Study Completion 2020-06 (Estimated)

PRIMARY OUTCOMES:
Postoperative Pain Score | day 1 postoperatively
  Visual analogue scale (0-5)

SECONDARY OUTCOMES:
Patient and parent satisfaction | Day 1 postoperatively
  Questionnaire: regarding how satisfied parents/ patients were with the treatment (satisfied or unsatisfied)
Quality of sleep | Day 1 post operative
  Questionnaire: (scale Child slept very well, average night sleep, poor nights sleep)
Postoperative Nausea and Vomiting | 4 hours postoperatively
  Questionnaire: vomiting, felt very nauseated, some nausea, none

CONTACTS AND LOCATIONS:
Locations (1):
- IWK Health Centre, Halifax, Nova Scotia, Canada

IPD SHARING:
Plan to Share IPD: No